CLINICAL TRIAL: NCT00580463
Title: Collection of Tumor Tissue, Blood and Spinal Fluid From Patients With Brain or Spine Tumors
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Rockefeller University (Other)
Responsible Party: Philip Gutin, MD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 99-125
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Primary or Metastatic Central Nervous System (CNS) Tumor
Keywords: central nervous system (CNS) tumor; tissue collection
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Spinal fluid

SUMMARY:
The purpose of the study is to collect samples of brain or spine tumors. Memorial Sloan-Kettering Cancer Center would then store them for use by researchers who study brain or spine cancer and try to find better ways of treating it. We will also collect blood and spinal fluid from patients with brain or spine tumors. The blood and spinal fluids are also used for research studies of cancer and its treatment.

DETAILED DESCRIPTION:
The main objective of the protocol is the establishment of a repository of central nervous system (CNS) tumors or metastases to the CNS and related tissues as an invaluable resource for current or future research studies of the etiology, pathogenesis and treatment of human central nervous system tumors. The database will be established through the intra-operative acquisition of brain or spine tumors as well as the collection of blood and spinal fluids from consenting CNS tumor patients.

ELIGIBILITY:
Inclusion Criteria:

* For acquisition of intra-operative brain or spine tumor specimens, blood specimens and spinal fluid specimens, all patients who undergo surgery for resection or biopsy qualify for inclusion in this protocol.
* If spinal fluid is not accessed as part of the operative procedure, it will not be collected.
* All patients must be under the care of one or more members of the MSKCC CNS disease management team at the time of tissue acquisition. Patients may have been previously diagnosed and/or treated at another institution.
* Subjects are eligible regardless of sex, age or race.
* Parental or guardian consents will be obtained in the case of minors (less than 18 years of age)

Exclusion Criteria:

* Patients or their guardians, in case of a minor, may choose to be excluded at any time.
* If a patient, or guardian, decides to withdraw after some or all of the tissues have been collected, such tissues will be destroyed at their request.
* Patients or their guardians will be counseled at the time of obtaining their consent, of the possibility of withdrawing from the protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient population will include adult and pediatric patients diagnosed with a primary or metastatic central nervous system tumor.
Sampling Method: Non-Probability Sample
Enrollment: 1128 (Actual)
Dates: Start 2000-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To establish a repository of CNS tumors or metastases to the CNS and related tissues for current or future studies. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gutin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org